CLINICAL TRIAL: NCT03745534
Title: Cochlear Implantation After Gamma Knife Radiosurgery with EABR and Correlation to Postoperative Hearing Results - a Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Christoph Arnoldner (Other)
Responsible Party: Sponsor-Investigator, Christoph Arnoldner, Assoc Prof PD. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 1564/2018
Record Dates: First submitted 2018-11-03; First posted 2018-11-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Vestibular Schwannoma; Hearing Loss
MeSH Terms: conditions — Neuroma, Acoustic; Hearing Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: eABR — eABR

SUMMARY:
Patients undergoing cochlear implantation after radio surgery for vestibular schwannoma will be included in the study. Patients will undergo preoperative and intraoperative eABR measurement. Correlations to postoperative hearing results will be drawn.

DETAILED DESCRIPTION:
Patients treated with radio surgery for vestibular schwannoma often suffer from hearing loss. Especially when the contralateral side has progressive hearing loss assessment if cochlear implantation is feasible, should be carried out. Patients undergo extensive audiometric testing. Additionally, patients will undergo preoperative eABR. Intraoperatively eABR is carried out and cochlear implantation is performed. The eABR results will be correlated with postoperative hearing. EABR measurements are not part of the study. The results of eBAR will be categorized in three groups (good response, weak response and no response). The eABR results will then be correlated to speech understanding with cochlear implants measured with Freiburger monosyllables test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone radio surgery for vestibular schwannoma
* Patients wanting cochlear implantation for hearing rehabilitation

Exclusion Criteria:

* Patients not wanting to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after radio surgery for vestibular schwannoma undergoing cochlear implantation
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
eABR correlation | 2 years
  eABR is correlated with postoperative hearing results eABR will be divided in three categories - good response, weak response, no response Hearing results will be measured with speech understanding in Freiburg monosyllables word test which is measured in % of monosyllables understanding at 65 and 80dB

CONTACTS AND LOCATIONS:
Locations (1):
- AKH; MUW, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No